CLINICAL TRIAL: NCT01297634
Title: Phase IV Study of Radial Diffusion of the Botulinum Toxin Type A: Electromyographic Evaluation of the Frontal Muscle.
Brief Title: Radial Diffusion of the Botulinum Toxin Type A (Botox®): Electromyographic Evaluation of the Frontal Muscle
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ivo Pitanguy Institute (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Armando Iniguez MD, Plastic Surgeon, Ivo Pitanguy Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 191622; 396936 (Other: CEP00/11); CEP001/11 (Other: Research Ethics Committee, Brazil)
Record Dates: First submitted 2011-02-16; First posted 2011-02-17 (Estimated); Last update posted 2011-11-23 (Estimated); Status verified 2011-11

CONDITIONS: Wrinkles
Keywords: Botulinum toxin type A; Hyperfunctional forehead lines; Randomized controlled trial; Double-blinded trial; Electromyogram (EMG); Electromyographic activity; Frontal Area
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Botulinum Toxin Type-A 1U (Other)
  Interventions: Drug: Botulinum Toxin Type-A (day 0)
- Botulinum Toxin Type-A 2U (Other)
  Interventions: Drug: Botulinum Toxin Type-A (day 0)
- Botulinum Toxin Type-A 3U (Other)
  Interventions: Drug: Botulinum Toxin Type-A (day 0)

INTERVENTIONS:
Drug: Botulinum Toxin Type-A (day 0) — * Botulinum Toxin Type-A 1 unit. Dilution:1U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 1 unit. Dilution: 0,5U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 1 unit. Dilution: 0,25U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  Arms: Botulinum Toxin Type-A 1U
Drug: Botulinum Toxin Type-A (day 0) — * Botulinum Toxin Type-A 2 Units. Dilution:1U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 2 units. Dilution: 0,5U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 2 units. Dilution: 0,25U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  Arms: Botulinum Toxin Type-A 2U
Drug: Botulinum Toxin Type-A (day 0) — Botulinum Toxin Type-A 3 units. Dilution:1U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 3 units. Dilution: 0,5U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  * Botulinum Toxin Type-A 3 units. Dilution: 0,25U/0,01ml (with saline solution). will be injected in the left and right belly to the Frontal Muscle.
  Arms: Botulinum Toxin Type-A 3U

SUMMARY:
This study evaluates the diffusion area (cephalic, lateral, medial and caudal points) of the botulinum toxin type A in the frontal muscle for usual concentrations and dilutions of the drug. A basal line control and After the application control will be made, and the investigators will evaluate the drug effects, based on clinical aspects, photographic registers and through electromyography exam (EMG).

Considering the results of our investigation, the investigators may propose a pattern of application of BOTULINUM TOXIN TYPE-A Botox® in the frontal area.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have indication for aesthetic treatment of the frontal dynamic wrinkles, in maximal contraction of the frontal muscle.
* Availability and understanding of the patient, for complete all the steps throughout the duration of the study.
* Medical history and physical examination compatible with the study.
* Informed consent signed.

Exclusion Criteria:

* Subjects with previous forehead face lifting or blepharoplasty surgery.
* Previous use of Botulinum toxin in the last 6 months.
* Forehead or eyelid asymmetry.
* Subjects with infections on site of injection or inflammatory skin diseases.
* Subjects with hypersensitivity to any component of the formulation, including albumin.
* Subjects with neuropathic or neuromuscular diseases.
* Subjects using aminoglycosides, penicillamine antibiotics, quinine and Ca2+ channel blockers.
* Subjects with pregnancy and lactation, or that planning become pregnant during the time of the study.
* Subjects with dimorphism or others psychological disorders.

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2011-05; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Treatment Area | Change from baseline at day 30
  Radial area (cephalic, lateral, medial and caudal points) of physioelectric activity of the frontal muscle, measured with electromyography (EMG).
  Clinical and Photographical register evaluation of the dynamical wrinkles in the treatment area.

SECONDARY OUTCOMES:
Complete Treatment Phase | Day 30
  Quantity of Botulinum Toxin used in every subject to aim to complete the treatment to the rest of the frontal area, based on the results of the primary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ivo Pitanguy Institute, Rio de Janeiro, Rio de Janeiro, Brazil